CLINICAL TRIAL: NCT03609268
Title: Effects of Stereotactic Body Radiotherapy and Microwave Ablation for Recurrent Small Hepatocellular Carcinoma: a Prospective, Randomized Controlled Study
Brief Title: Stereotactic Body Radiotherapy and Microwave Ablation for Recurrent Small Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR2018001025
Record Dates: First submitted 2018-07-02; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Recurrent Hepatocellular Carcinoma; Microwave Ablation; Stereotactic Body Radiotherapy
Keywords: Recurrent Hepatocellular Carcinoma; Microwave ablation; Stereotactic body radiotherapy; Small liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MWA (Active Comparator): Patients receive microwave ablation (MWA)
  Interventions: Device: microwave ablation (MWA)
- SBRT (Experimental): Patients receive stereotactic body radiotherapy (SBRT)
  Interventions: Radiation: stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Device: microwave ablation (MWA) — microwave ablation (MWA) for recurrent small liver cancer
  Arms: MWA
Radiation: stereotactic body radiotherapy (SBRT) — stereotactic body radiotherapy (SBRT) for recurrent small liver cancer
  Arms: SBRT

SUMMARY:
The prognosis of small liver cancer (≤5 cm) who had underwent stereotactic body radiotherapy (SBRT) is encouraging, with the 1-year local control rate has been reported to be 95-100%, 3-year local control rate about 91%, 3-year overall survival rate around 70%. Local ablation therapy has become the standard treatment for recurrent liver cancer after surgery and interventional treatment. The ablation rate of tumors with a diameter of 3.1-5.0 cm reached 90%. The 1, 2, and 3-year survival rates had been reported to be 89%, 74%, and 60%, respectively, which is similar to that of surgical resection. At present, there is no randomized controlled study of SBRT and microwave ablation (MWA) for small liver cancer. It is hoped that this study will further compare the efficacy of SBRT and MWA for recurrent small hepatocellular carcinoma.

DETAILED DESCRIPTION:
Recurrent small hepatocellular carcinoma after surgery or local ablation therapy are chose for this study. The patients are divided into two groups randomly. Patients in group A receive MWA, group B patients receive SBRT. The 3-year progression free survival, 3-year local recurrence free survival, 3-year overall survival and other endpoints events were recorded and analyzed, to assess whether SBRT is non-inferior to MWA.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old and above.
2. Clinical or pathological diagnosis of recurrent hepatocellular carcinoma after initial treatment (surgery, TACE, radiofrequency ablation, etc.)
3. Small hepatocellular carcinoma meeting the Milan criteria: single lesion ≤ 5cm, or tumor number ≤ 3, maximum diameter ≤ 3cm, no major vascular invasion of portal vein, hepatic vein, inferior vena cava, no bile duct invasion, no lymph node and extrahepatic metastasis
4. No serious blood system, heart, lung, liver, kidney dysfunction and immune deficiency
5. The neutrophil count is at least 1.0*10^9/ml, and the platelet count is at least 50*10^9/ml. Hemoglobin is at least 80g/L.
6. Men or women with fertility are willing to take contraceptive measures during the trial
7. Eastern Cooperative Oncology Group score 0-1 points
8. Expected survival period > 3 months
9. Voluntary participation and signing of informed consent

Exclusion Criteria:

1. Patients who have undergone chemoradiation or targeted therapy for liver cancer
2. Obvious cirrhosis, recent hematemesis due to portal hypertension, Child-Pugh score ≥10 points
3. Total bilirubin >70umol/L, aspartate aminotransferase (ALT), alanine aminotransferase (AST) exceed the upper limit of normal 3 times.
4. Patients undergoing major surgery within 1 month of study initiation
5. Patients with previous history of malignancy (excludes tumor-free survival after treatment of basal cell carcinoma of the skin and carcinoma of the cervix in situ for more than 3 years)
6. Researchers consider it inappropriate to participate in the test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-06-30 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
progression free survival | From the date of MWA or the first fraction of SBRT until the date of first progression (local or distant), assessed up to 3 years.
  Progression-free survival (PFS) was measured from the date of MWA or the first fraction of SBRT until the date of first progression (local or distant).

SECONDARY OUTCOMES:
local recurrence free survival | From the date of MWA or the first fraction of SBRT until the date of local recurrence, assessed up to 3 years
  Local recurrence free survival (LRFS) was measured from the date of MWA or the first fraction of SBRT until the date of local recurrence.
overall survival | From the date of MWA or the first fraction of SBRT until the date of death, assessed up to 3 years
  Overall survival (OS) was measured from the date of MWA or the first fraction of SBRT until the date of death.

CONTACTS AND LOCATIONS:
Locations (1):
- the second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China